CLINICAL TRIAL: NCT03619486
Title: Low Energy Shock Wave for the Treatment of Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) - a Randomized, Double-blind, Placebo-controlled, Prospective Study
Brief Title: Low Energy Shock Wave for the Treatment of Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201800525A3
Record Dates: First submitted 2018-07-19; First posted 2018-08-08 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Interstitial Cystitis
Keywords: Low Energy Shock Wave (LESW); Extracorporeal Shockwave Therapy; interstitial cystitis/bladder pain syndrome (IC/BPS)
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: Double blind, placebo control study. Eligible participants will be assigned a randomization number in sequential order and each of the randomization will determine the allocation of one of the two treatment groups (LESW and Placebo) in 1: 1 ratio as shown below. The LESW and placebo will be controlled by a research assistance who will not evaluate the therapeutic outcome to ensure the double blind method.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo treatment (shock wave probe w/o energy)
  Interventions: Device: Placebo
- Low energy shock wave (Experimental): Low energy shock wave treatment (shock wave probe w/ energy)
  Interventions: Device: Low energy shock wave

INTERVENTIONS:
Device: Low energy shock wave — Probe be transcutaneous applied to the suprapubic bladder region with 2000 shocks, frequency of 3 pulses per second and maximum total energy flow density 0.25 millijoule/mm2 once a week for 4 weeks
  Arms: Low energy shock wave
Device: Placebo — Probe be transcutaneous applied to the suprapubic bladder region with 2000 shocks, frequency of 3 pulses per second but no energy once a week for 4 weeks
  Arms: Placebo

SUMMARY:
To investigate the efficacy and safety of LESW on participants with IC/BPS

DETAILED DESCRIPTION:
Low energy shock wave (LESW) is known to facilitate tissue regeneration with analgesic and anti-inflammatory effects. LESW has been proved to have therapeutic effects in patients with nonbacterial prostatitis and chronic pelvic pain syndrome (CPPS). Investigator's previous study has demonstrated that LESW treatment inhibited nerve growth factor (NGF), interleukin-6 (IL-6), and cyclooxygenase-2 (COX-2) expression, and blocked the bladder pain, inflammation and overactivity in a cyclophosphamide induced cystitis model in rats. These findings suggest that a potential clinical benefit of LESW treatment for patients with interstitial cystitis/bladder pain syndrome (IC/BPS).

A total of 50 participants with IC/BPS will be enrolled to receive LESW (transcutaneous applied to the suprapubic bladder region with 2000 shocks, frequency of 3 pulses per second and maximum total energy flow density 0.25 millijoule/mm2) once a week for 4 weeks or placebo (same condition but with no energy) treatment.

All participants should have IC symptoms for at least 6 months, and have received cystoscopy to rule out other bladder lesion. Participants should not have urinary tract infection (UTI) in recent 3 months, and no urinary tract stone. Participants should not receive intravesical hyaluronic acid treatment in recent 3 months, or intravesical Botox injection in recent 12 months. Retreatment with LESW at 3 months if participants reports ineffective.

Primary end-point is the change of the O'Leary-Sant symptom score (OSS), including Interstitial Cystitis Symptom Index (ICSI) and Interstitial Cystitis Problem Index (ICPI) from baseline to 1 month after treatment. Secondary endpoints include Visual Analogue Scale (VAS), daily frequency, nocturia and functional bladder capacity (FBC) as record in 3-day voiding diary, maximum flow rate (Qmax), voided volume, postvoiding residual (PVR) and global response assessment (GRA). Two visits are required at baseline screening (before first treatment), treatment (V1), 1 week (V2), 2 weeks (V3), 3 weeks (V4) and 1 week post V4 treatment (V5), 1 month post V4 treatment (V6, primary end-point), and 3 months post V4 treatment (V7) . Urine samples will be collected at each time-point for NGF and cytokines tests. Bladder biopsy will be performed at baseline and repeat cystoscopy at 3 months post treatment optional.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with age of 20 years old or above
2. Patients with symptoms of unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms of more than six months duration, in the absence of infection or other identifiable causes
3. Patients has received cystoscopy and ruled out other bladder lesion
4. Free of active urinary tract infection
5. Free of bladder outlet obstruction on enrollment
6. Free of overt neurogenic bladder dysfunction and limitation of ambulation
7. Patient or his/her legally acceptable representative has signed the written informed consent form

Exclusion Criteria:

1. Patients had received intravesical hyaluronic acid treatment in recent 3 months, or intravesical Botox injection in recent 12 months Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
2. Patients with bladder outlet obstruction on enrollment
3. Patients with PVR >100 ml
4. Patients with uncontrolled confirmed diagnosis of acute urinary tract infection
5. Patients have laboratory abnormalities at screening including: alanine aminotransferase (ALT)> 3 x upper limit of normal range, and aspartate aminotransferase (AST) > 3 x upper limit of normal range
6. Patients have abnormal serum creatinine level > 2 x upper limit of normal range
7. Female patients who is pregnant, lactating, or with child-bearing potential without contraception
8. Patients with any other serious disease considered by the investigator not in the condition to enter the trial
9. Patients had received intravesical treatment for IC within recent 1 month
10. Patients had participated investigational drug trial within 1 month before entering this study
11. Patients with coagulopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change of the O'Leary-Sant symptom score (OSS, including ICSI and ICPI) | Baseline and 1 month
  Change of the O'Leary-Sant symptom score from baseline to 1 month after the treatment day.
  Subscales ICSI and ICPI are graded from 0 to 20 and 0 to 16, respectively. The items are summed to obtain OSS (range from 0 to 36, higher values represent a worse outcome).

SECONDARY OUTCOMES:
Net changes of the Visual Analog Scale (VAS) | Baseline and 1 month
  Net changes of the Visual Analog Scale from baseline to 1 month after the treatment day (VAS range from 0 to 10, higher values represent a worse outcome)
Net changes of the functional bladder capacity (FBC) as assessed by the maximum urine volume (milliliters) as recorded in 3-day voiding diary | Baseline and 1 month
  Net changes of the functional bladder capacity (FBC) from baseline to 1 month after the treatment day (higher FBC volumes represent a better outcome)
Net changes of the voiding frequency at daytime as recorded in 3-day voiding diary | Baseline and 1 month
  Net changes of the voiding frequency at daytime as recorded in 3-day voiding diary from baseline to 1 month after the treatment day (higher voiding frequency at daytime represent a worse outcome)
Net changes of the voiding frequency at night time as recorded in 3-day voiding diary | Baseline and 1 month
  Net changes of the voiding frequency at night time as recorded in 3-day voiding diary from baseline to 1 month after the treatment day (higher voiding frequency at night time represent a worse outcome)
Net changes of the Global response assessment (GRA) | Baseline and 3 month
  Global response assessment (GRA) of therapeutic result by the patient (categorized from -3 to +3, indicating markedly worse to markedly improved) at 3 months after the last treatment day
Net changes of the maximum flow rate | Baseline and 1 month
  Net changes of the maximum flow rate from baseline to 1 month after the treatment day (higher maximum flow rate represent a better outcome)
Net changes of the voided volume | Baseline and 1 month
  Net changes of the voided volume from baseline to 1 month after the treatment day (higher voided volumes represent a better outcome)
Net changes of the PVR | Baseline and 1 month
  Net changes of the PVR from baseline to 1 month after the treatment day (higher PVR volumes represent a worse outcome)
Net changes of the cytokines level | Baseline and 1 month
  Net changes of the cytokines level from baseline to 1 month after the treatment day (e.g. NGF and IL-6, higher values represent a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang Hsieh, MD, Study Chair — Institutional Review Board Chang Gung Medical Foundation
Locations (1):
- Chang Gung Memorial Hospital, Chang Gung University College of Medicine, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Hanno PM, Burks DA, Clemens JQ, Dmochowski RR, Erickson D, Fitzgerald MP, Forrest JB, Gordon B, Gray M, Mayer RD, Newman D, Nyberg L Jr, Payne CK, Wesselmann U, Faraday MM; Interstitial Cystitis Guidelines Panel of the American Urological Association Education and Research, Inc. AUA guideline for the diagnosis and treatment of interstitial cystitis/bladder pain syndrome. J Urol. 2011 Jun;185(6):2162-70. doi: 10.1016/j.juro.2011.03.064. Epub 2011 Apr 16. PMID 21497847
- [Background] Hanno PM, Sant GR. Clinical highlights of the National Institute of Diabetes and Digestive and Kidney Diseases/Interstitial Cystitis Association scientific conference on interstitial cystitis. Urology. 2001 Jun;57(6 Suppl 1):2-6. doi: 10.1016/s0090-4295(01)01112-8. PMID 11378041
- [Background] Nickel JC, Barkin J, Forrest J, Mosbaugh PG, Hernandez-Graulau J, Kaufman D, Lloyd K, Evans RJ, Parsons CL, Atkinson LE; Elmiron Study Group. Randomized, double-blind, dose-ranging study of pentosan polysulfate sodium for interstitial cystitis. Urology. 2005 Apr;65(4):654-8. doi: 10.1016/j.urology.2004.10.071. PMID 15833501
- [Background] Hanno PM, Buehler J, Wein AJ. Use of amitriptyline in the treatment of interstitial cystitis. J Urol. 1989 Apr;141(4):846-8. doi: 10.1016/s0022-5347(17)41029-9. PMID 2926877
- [Background] Sairanen J, Forsell T, Ruutu M. Long-term outcome of patients with interstitial cystitis treated with low dose cyclosporine A. J Urol. 2004 Jun;171(6 Pt 1):2138-41. doi: 10.1097/01.ju.0000125139.91203.7a. PMID 15126772
- [Background] Hanno PM, Erickson D, Moldwin R, Faraday MM; American Urological Association. Diagnosis and treatment of interstitial cystitis/bladder pain syndrome: AUA guideline amendment. J Urol. 2015 May;193(5):1545-53. doi: 10.1016/j.juro.2015.01.086. Epub 2015 Jan 23. PMID 25623737
- [Background] Chancellor MB, Yoshimura N. Treatment of interstitial cystitis. Urology. 2004 Mar;63(3 Suppl 1):85-92. doi: 10.1016/j.urology.2003.10.034. PMID 15013658
- [Background] Shie JH, Liu HT, Kuo HC. Increased cell apoptosis of urothelium mediated by inflammation in interstitial cystitis/painful bladder syndrome. Urology. 2012 Feb;79(2):484.e7-13. doi: 10.1016/j.urology.2011.09.049. PMID 22310775
- [Background] Lee JD, Lee MH. Increased expression of hypoxia-inducible factor-1alpha and vascular endothelial growth factor associated with glomerulation formation in patients with interstitial cystitis. Urology. 2011 Oct;78(4):971.e11-5. doi: 10.1016/j.urology.2011.05.050. Epub 2011 Aug 2. PMID 21813166
- [Background] Chaussy C, Schmiedt E, Jocham D, Brendel W, Forssmann B, Walther V. First clinical experience with extracorporeally induced destruction of kidney stones by shock waves. J Urol. 1982 Mar;127(3):417-20. doi: 10.1016/s0022-5347(17)53841-0. PMID 6977650
- [Background] Wang CJ. An overview of shock wave therapy in musculoskeletal disorders. Chang Gung Med J. 2003 Apr;26(4):220-32. PMID 12846521
- [Background] Di Meglio F, Nurzynska D, Castaldo C, Miraglia R, Romano V, De Angelis A, Piegari E, Russo S, Montagnani S. Cardiac shock wave therapy: assessment of safety and new insights into mechanisms of tissue regeneration. J Cell Mol Med. 2012 Apr;16(4):936-42. doi: 10.1111/j.1582-4934.2011.01393.x. PMID 21790971
- [Background] Vardi Y, Appel B, Kilchevsky A, Gruenwald I. Does low intensity extracorporeal shock wave therapy have a physiological effect on erectile function? Short-term results of a randomized, double-blind, sham controlled study. J Urol. 2012 May;187(5):1769-75. doi: 10.1016/j.juro.2011.12.117. Epub 2012 Mar 15. PMID 22425129
- [Background] Mariotto S, de Prati AC, Cavalieri E, Amelio E, Marlinghaus E, Suzuki H. Extracorporeal shock wave therapy in inflammatory diseases: molecular mechanism that triggers anti-inflammatory action. Curr Med Chem. 2009;16(19):2366-72. doi: 10.2174/092986709788682119. PMID 19601786
- [Background] Wang HJ, Lee WC, Tyagi P, Huang CC, Chuang YC. Effects of low energy shock wave therapy on inflammatory moleculars, bladder pain, and bladder function in a rat cystitis model. Neurourol Urodyn. 2017 Aug;36(6):1440-1447. doi: 10.1002/nau.23141. Epub 2016 Dec 30. PMID 28035695
- [Background] Zimmermann R, Cumpanas A, Miclea F, Janetschek G. Extracorporeal shock wave therapy for the treatment of chronic pelvic pain syndrome in males: a randomised, double-blind, placebo-controlled study. Eur Urol. 2009 Sep;56(3):418-24. doi: 10.1016/j.eururo.2009.03.043. Epub 2009 Mar 25. PMID 19372000
- [Background] Al Edwan GM, Muheilan MM, Atta ON. Long term efficacy of extracorporeal shock wave therapy [ESWT] for treatment of refractory chronic abacterial prostatitis. Ann Med Surg (Lond). 2017 Jan 6;14:12-17. doi: 10.1016/j.amsu.2016.12.051. eCollection 2017 Feb. PMID 28119778
- [Result] Chuang YC, Meng E, Chancellor M, Kuo HC. Pain reduction realized with extracorporeal shock wave therapy for the treatment of symptoms associated with interstitial cystitis/bladder pain syndrome-A prospective, multicenter, randomized, double-blind, placebo-controlled study. Neurourol Urodyn. 2020 Jun;39(5):1505-1514. doi: 10.1002/nau.24382. Epub 2020 May 11. PMID 32394478
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

DOCUMENTS (2):
  • Study Protocol (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT03619486/Prot_002.pdf
  • Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT03619486/SAP_003.pdf